CLINICAL TRIAL: NCT06290934
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose-Ranging Study Evaluating the Efficacy and Safety of GS-1427 in Adult Participants With Moderately to Severely Active Ulcerative Colitis (UC)
Brief Title: Study of GS-1427 in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: SWIFT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-409-5704; 2023-508304-38 (Other: European Medicines Agency)
Record Dates: First submitted 2024-02-16; First posted 2024-03-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A, Part B, Part C: GS-1427 Dose A (Experimental): Participants will receive GS-1427 Dose A Day 1 through Week 12 (Part A).
  Participants who complete the 12-week Part A treatment period will be eligible to continue and remain on the same dose of GS-1427 through Week 52 (Part B).
  Participants who complete Part B of the study will continue onto Part C: Blinded treatment extension for an additional 24 weeks (through Week 76).
  Interventions: Drug: GS-1427
- Part A, Part B, Part C: GS-1427 Dose B (Experimental): Participants will receive GS-1427 Dose B Day 1 through Week 12 (Part A).
  Participants who complete the 12-week Part A treatment period will be eligible to continue and remain on the same dose of GS-1427 through Week 52 (Part B).
  Participants who complete Part B of the study will continue onto Part C: Blinded treatment extension for an additional 24 weeks (through Week 76).
  Interventions: Drug: GS-1427
- Part A, Part B, Part C: GS-1427 Dose C (Experimental): Participants will receive GS-1427 Dose C Day 1 through Week 12 (Part A).
  Participants who complete the 12-week Part A treatment period will be eligible to continue and remain on the same dose of GS-1427 through Week 52 (Part B).
  Participants who complete Part B of the study will continue onto Part C: blinded treatment extension for an additional 24 weeks (through Week 76).
  Interventions: Drug: GS-1427
- Part A, Placebo; Part B, Part C: GS-1427 (Experimental): Participants will receive Placebo to match GS-1427 Day 1 through Week 12 (Part A). Part A placebo participants will be eligible to undergo re-randomization in a double-blind manner after endoscopy assessment at Week 12 to receive one of the GS-1427 dose A, B, or C treatments.
  Participants will be eligible to continue and remain on the new dose through Week 52 (Part B). Participants who complete Part B of the study will continue onto Part C: blinded treatment extension for an additional 24 weeks (through Week 76).
  Interventions: Drug: GS-1427; Drug: Placebo-to-match GS-1427

INTERVENTIONS:
Drug: GS-1427 — Administered orally
Drug: Placebo-to-match GS-1427 — Administered orally
  Arms: Part A, Placebo; Part B, Part C: GS-1427

SUMMARY:
The goal of this study is to learn if GS-1427 is effective in treating participants with moderate to severe ulcerative colitis. The study will compare participants in different treatment groups treated with GS-1427 with participants treated with placebo.

The primary objective of this study is to assess the efficacy of GS-1427, compared with placebo control, in achieving clinical response at Week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals have Ulcerative Colitis (UC) with symptoms of at least 90 days duration before randomization, with the diagnosis confirmed by endoscopy and histology at any time prior to randomization. Documentation of endoscopy and histology consistent with the diagnosis of UC must be available in the source documents.
* Individuals have UC with minimum disease extent of 15 cm from the anal verge.
* Individuals have moderately to severely active UC as determined by endoscopy occurring during screening with a total modified Mayo Clinic Score (mMCS) of 5 to 9 points, including a centrally read endoscopic subscore of at least 2.
* Individuals have an inadequate response or loss of response or are intolerant to at least 1 of the following UC treatments: corticosteroids, immunomodulators, or advanced therapy.
* Individuals have an inadequate response or loss of response or are intolerant to < 3 AT mechanisms of action for UC (use of 2 or more AT with the same mechanism of action, eg, 2 TNF-α inhibitors, counts as 1 mechanism of action)

Key Exclusion Criteria:

* Have a current diagnosis of Crohn's Disease (CD) or clinical findings suggestive of CD, diagnosis of indeterminate colitis due to etiologies such as an enteric pathogen, or lymphocytic or collagenous colitis.
* Have a current diagnosis of toxic megacolon, symptomatic colonic stricture, acute severe colitis, fulminant colitis, or abdominal abscess at screening or randomization.
* Have any history of exposure to vedolizumab or other integrin antagonists
* Requirement for ongoing therapy with or use of any prohibited medication as specified in the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Clinical Response at Week 12 | Week 12
  Clinical response is defined as a decrease from baseline in the modified Mayo Clinic Score (mMCS) of ≥ 2 points and at least a 30% reduction from baseline, and a decrease in rectal bleeding subscore of ≥ 1 from baseline or an absolute rectal bleeding subscore of 0 or 1. The mMCS is a scoring system for assessment of Ulcerative Colitis (UC) activity and is composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease (spontaneous bleeding, ulceration)), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), and stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 or more stools more than normal). Total score for mMCS ranges from 0 to 9 (sum of all subscores), with higher scores indicating higher disease activity.

SECONDARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), or Deaths. | First dose date up to 76 weeks plus 28 days
Incidence of Treatment-emergent Lab Abnormalities | First dose date up to 76 weeks plus 28 days
Proportion of Participants Achieving Clinical Remission at Week 12 | Week 12
  Clinical remission is defined as a mMCS of ≤ 2, including a stool frequency subscore (SFS) ≤ 1 and not greater than baseline, rectal bleeding subscore of 0, and centrally read endoscopic subscore ≤ 1 (score of 1 modified to exclude friability).The mMCS is a scoring system for assessment of UC activity and is composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease (spontaneous bleeding, ulceration)), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), and stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 or more stools more than normal). Total score for mMCS ranges from 0 to 9 (sum of all subscores), with higher scores indicating higher disease activity.
Proportion of Participants Achieving Clinical Remission at Week 52 | Week 52
  Clinical remission is defined as a mMCS of ≤ 2, including a stool frequency subscore (SFS) ≤ 1 and not greater than baseline, rectal bleeding subscore of 0, and centrally read endoscopic subscore ≤ 1 (score of 1 modified to exclude friability). The mMCS is a scoring system for assessment of UC activity and is composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease (spontaneous bleeding, ulceration)), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), and stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 or more stools more than normal). Total score for mMCS ranges from 0 to 9 (sum of all subscores), with higher scores indicating higher disease activity.
Proportion of Participants Achieving Histologic-endoscopic Mucosal Improvement at Week 12 | Week 12
  Histologic-endoscopic mucosal improvement is a composite endpoint that uses different units of measure for histologic and endoscopic activities.Histologic activity is measured by the Geboes score with 6 grades:0,structural change(sub-grade:0.0-0.3);1,chronic inflammatory infiltrate(sub-grade:1.0-1.3);2,lamina propria neutrophils & eosinophils(sub-grade:2A.0-2B.3);3,neutrophils in epithelium(sub-grade:3.0-3.3);4,crypt destruction(sub-grade:4.0-4.3); and 5,erosion or ulceration(sub-grade:5.0-5.4);final score range 0.0-5.4;higher scores indicate more severe inflammation.Endoscopic activity is measured by the Mayo Clinic Score Endoscopic subscores(range 0-3):0,normal or inactive disease;1,mild disease(erythema,decreased vascular pattern);2,moderate disease(marked erythema,lack of vascular pattern,friability,erosions), and 3,severe disease(spontaneous bleeding,ulceration).Histologic-endoscopic mucosal improvement is defined as achieving both Geboes score ≤ 3.1 and endoscopic subscore ≤ 1
Proportion of Participants Achieving Mucosal Healing at Week 12 | Week 12
  Mucosal healing is a composite endpoint that uses different units of measure for histologic and endoscopic activities. Histologic activity is measured by the Geboes score with 6 grades:0,structural change(sub-grade:0.0-0.3);1,chronic inflammatory infiltrate(sub-grade:1.0-1.3);2,lamina propria neutrophils & eosinophils(sub-grade:2A.0-2B.3);3,neutrophils in epithelium(sub-grade:3.0-3.3);4,crypt destruction(sub-grade:4.0-4.3); and 5,erosion or ulceration(sub-grade:5.0-5.4);final score range 0.0-5.4;higher scores indicate more severe inflammation.Endoscopic activity is measured by the Mayo Clinic Score Endoscopic subscores(range 0-3):0,normal or inactive disease;1,mild disease(erythema,decreased vascular pattern);2,moderate disease(marked erythema,lack of vascular pattern,friability,erosions), and 3,severe disease(spontaneous bleeding,ulceration).Mucosal healing is defined as achieving both Geboes score ≤ 2B.1 and endoscopic subscore ≤ 1.
Proportion of Participants Achieving Endoscopic Improvement at Week 12 | Week 12
  Endoscopic improvement is defined as an endoscopic subscore of ≤ 1. Endoscopic subscore is a part of the modified Mayo Clinic Score which is a scoring system for assessment of UC activity. Endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern), 2 = moderate disease (marked erythema, lack of vascular pattern, friability, erosions), and 3 = severe disease (spontaneous bleeding, ulceration).
To Assess the Efficacy of GS-1427 in Achieving Partial Modified Mayo Clinic Score (mMCS) remission at Week 76 | Week 76

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (181):
- United States (56):
  - Onyx Clinical Research (Clinic Location), Peoria, Arizona
  - Om Research LLC, Camarillo, California
  - VVCRD Research, Garden Grove, California
  - 310 Clinical Research, Inglewood, California
  - US San Diego Health System, La Jolla, California
  - Om Research LLC, Lancaster, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University Of California, Davis, Sacramento, California
  - SDG Clinical Research, LLC, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Gastro Florida, Clearwater, Florida
  - Best Quality Research, Inc, Hialeah, Florida
  - United Research Institute LLC, Hialeah, Florida
  - University of Miami Hospital and Clinics, Sylvester Comprehensive Cancer Center(Drug shipment)-Research Pharmacy, Miami, Florida
  - Medical Professional Clinical Research Center, Inc., Miami, Florida
  - Blessed Health Care & Research, Inc, Miami, Florida
  - Alliance Clinical Research of Tampa, LLC, New Port Richey, Florida
  - Digestive and Liver Center of Florida, LLC, Orlando, Florida
  - Clinical Research of Osceola, Orlando, Florida
  - Encore Medical Research of Weston, LLC, Weston, Florida
  - EBGS Clinical Research Center, Snellville, Georgia
  - The University of Chicago Medical Center (Duchossois Center for Advanced Medicine), Chicago, Illinois
  - Onyx Clinical Research, Peoria, Illinois
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinical Research Center., Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Gastroenterology Associates of North Mississippi, Oxford, Mississippi
  - Digestive Health Specialists (Clinic Visits), Tupelo, Mississippi
  - St Charles Clinical Research, Weldon Spring, Missouri
  - Tandem - Allied Clinical Research, LLC, Freehold, New Jersey
  - N.Y. Total Medical Care, PC, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Lenox Hill Hospital, Manhasset, New York
  - NYU Grossman School of Medicne, New York, New York
  - Carolina Research, Greenville, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Dayton Gastroenterology, LLC, Beavercreek, Ohio
  - Gastro Health Research, Cincinnati, Ohio
  - NexGen Research, Lima, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio, LLC, Westlake, Ohio
  - Penn State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Skyline gastroenterology of west Tennessee, Jackson, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Vanderbilt Inflammatory Bowel Disease Clinic, Nashville, Tennessee
  - Gastroenterology Research of San Antonio, Fredericksburg, Texas
  - Amel Med Llc, Georgetown, Texas
  - GI Alliance - Mansfield, Mansfield, Texas
  - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Southern Star Research Institute, LLC., San Antonio, Texas
  - Tyler Research Institute, LLC., Tyler, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Emeritas Research Group, Lansdowne Town Center, Virginia
  - Gastroenterology Consultants of Southwest Virginia, Roanoke, Virginia
- Australia (8):
  - Macquarie University, Sydney, New South Wales
  - Mater Adult Hospital - Mater Misericordiae Ltd and Mater Research Ltd, South Brisbane, Queensland
  - Princess Alexandra Hospital - Metro South Health, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Monash Health - Monash Medical Centre, Clayton, Victoria
  - Northern Hospital - Northern Health, Epping, Victoria
  - Saint Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital - Westerm Health, Footscray, Victoria
- Austria (3):
  - Medical University Innsbruck, University Hospital for Internal Medicine I, Innsbruck
  - Regional Hospital Salzburg, University Clinic for Internal Medicine I, Salzburg
  - Medical University Vienna, Department of Internal Medicine Division Gastroenterology and Hepatology, Vienna
- Belgium (3):
  - Imeldaziekenhuis, Bonheiden
  - AZ Groeninge, Kortrijk
  - Vitaz, Sint-Niklaas
- TDDA Specialty Reserach, Vaughan, Canada
- Czechia (2):
  - PreventaMed, s.r.o., Olomouc
  - Nemocnice Slany, Slaný
- France (3):
  - Centre Hospitalier Universitaire Grenoble Alpes(CHUGA) - Service Hepato-Gastroentérologie, 7éme unité D, La Tronche
  - CHU Nantes Gastroenterology department, Nantes
  - Hospices Civilis de Lyon - Hospital Lyon Sud Department of Gastroenterology, Pierre-Bénite
- ARENSIA Exploratory Medicine, Tbilisi, Georgia
- Germany (4):
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Medizinische Klinik und Poliklinik |, Dresden
  - Studiengesellschaft BSF UG, Halle
  - University Hospital Schleswig-Holstein, Clinic for Internal Medicine, Kiel
  - Ulm University Hospital, Centre for Internal Medicine I, Ulm
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
- Hungary (4):
  - Békés Varmegye Kozponti Korhaz, dr Rethy Pal 4. Belgyégyaszat - Gasztroenterologia, Békéscsaba
  - Semmelweis Egyetem AOK, Budapest
  - Semmelweis Egyetem Általanos Orvostudományi Kar, Budapest
  - Clinexpert Gyógycentrum, Budapest
- Italy (12):
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS, Bologna
  - Azienda Ospedaliera Brotzu - P.O. San Michele, Cagliari
  - AOU "Renato Dulbecco" - Digestive Physiopathology Unit, Catanzaro
  - San Raffaele Hospital IRCCS, Milan
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar
  - Azienda Ospedale Universita di Padova, Padua
  - AOOR Villa Sofia- Cervello, Palermo
  - Campus Biomedico University Hospital Foundation, Roma
  - Ospedale Sandro Pertini, Roma
  - IRCCS Policlinico San Donato, San Donato Milanese
  - Ospedale Casa Sollievo della Sofferenza IRCCS, Opera di San Pio da Pietrelcina, San Giovanni Rotondo
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Malaysia (7):
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Universiti Sains Malaysia, Kelantan
  - Hospital Queen Elizabeth, Kota Kinabalu
  - Hospital Sultan Idris Shah Serdang, Kuala Selangor
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Sultan Ahmad Shah Medical Centre @IIUM, Kuantan
  - University Malaya Medical Centre, Petaling Jaya
- PMSI Clinical Republican Hospital "Timofei Molneaga", Chisinau, Moldova
- New Zealand (3):
  - Pacific Clinical Research Network - Auckland, Auckland
  - Christchurch Hospital, Christchurch
  - Health New Zealand - Te Whatu Ora Southern, Gastroenterology Department, Dunedin Hospital, Dunedin
- Poland (22):
  - Centrum Medyczne "Medis", Bydgoszcz
  - NZOZ Holsamed - Oddzial Libero, Katowice
  - Centrum Medyczne Plejady Magdalena Celinska Loewenhoff Michal Zolnowski sp.k., Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Ksawerów
  - Medrise Sp. z o.o., Lublin
  - Centrum Innowacyjnych Terapii Sp. z o.o., Mazowieckie
  - EMC Instytut Medyczny SA PL Certus Szpital Nr 1 PL Certus Ambulatorium, Poznan
  - Gabinety Lekarskie RIVERMED, Poznan
  - Centrum Medyczne Medyk Sp. z 0.0. sp.k., Rzeszów
  - Endoskopia Sp. z.o.o., Sopot
  - Sonomed Sp. z 0.0., Szczecin
  - Twoja Przychodnia Szczecinskie Centrum Medyczne Sp. zo.o., Szczecin
  - Gastromed Sp. z.o.o., Torun
  - H-T Centrum Medyczne - Endoterapia, Tychy
  - Bodyclinic Sp. z o.o. sp.k., Warsaw
  - Przychodnia care Access Warsawa, Warsaw
  - Medical Network Sp. z 0.0. WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej Vivamed Jadwiga Miecz, Warsaw
  - FutureMeds Wrocław, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - Przychodnia Euromedicare szpital euromedicare, Wroclaw
- Romania (11):
  - Spitalul Universitar De Urgenta Militar Central Dr. Carol Davila, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Centrul Medical Medicum S.R.L., Bucharest
  - Centrul Medical Monza S.R.L, Bucharest
  - Spitalul Clinic Judetean De Urgenta Cluj-Napoca, Cluj-Napoca
  - Institutul Regional De Gastroenterologie Hepatologie Prof. Dr. Octavian Fodor Cluj-Napoca, Cluj-Napoca
  - Gastromed S.R.L, Constanța
  - Spitalul Judetean de Urgenta Satu Mare, Satu Mare
  - Asociatia Oncohelp, Timișoara
  - Centrul De Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Serbia (6):
  - Clinical Hospital Center "Bezanijska Kosa", Clinic for Internal Medicine, Gastroenterology and Hepatology Department, Belgrade
  - Clinical Hospital Center "Dr Dragisa Misovic - Dedinje" Clinic for Intemal Medicine, Gastroentero logy and Hepatology Department, Belgrade
  - Clinical Hospital Center "Zvezdara" - Belgrade, Clinic for Internal Diseases Clinical Department of Gastroenterology and Hepatology, Belgrade
  - University Clinical Center of Serbia, Clinic for Gastroenterology and Hepatology, Belgrade
  - University Clinical Center Kragujevac, Clinic for Gastroenterology and Hepatology, Kragujevac
  - General Hospital "Djordje Joanovic" Zrenjanin,Internal Medicine Sector - Internal Department, Zrenjanin
- South Korea (12):
  - Inje University Haeundae Paik Hospital IRB, Busan
  - Kyungpook National University Hospital, Daegu
  - The Catholic University of Korea Daejeon St.Mary's Hospital, Daejeon
  - Kyung Hee University Hospital, Guri-si
  - Kangbuk Samsung Hospital, Jongno-Gu
  - Yeungnam University Hospital, Nam-Gu
  - Hanyang University Seoul Hospital, Seongdong-gu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (6):
  - Hospital Arquitecto Marcide. Complejo Hospitalario Universitario de Ferrol, Ferrol
  - Hospital Universitario de Cabuenes, Gijón
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario Nuestra Senora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, 7, Chung-Shan South Road, Taipei, ZIP 100, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital (CGMH), Taoyuan
- United Kingdom (6):
  - Southmead Hospital - North Bristol Trust Clinical Research Centre, Bristol
  - Fairfield General Hospital, Northerncare Alliance NHS Foundation Trust, Bury
  - Cambridge University Hospital NHS Trust, Addenbrookes Hospital, Cambridge
  - Synexus Clinical Research Centre, Cardiff
  - King's College Hospital, London
  - Northumbria Healthcare NHS Foundation Trust, North Tyneside General Hospital, North Shields

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06290934